CLINICAL TRIAL: NCT00524667
Title: HDAC Inhibitor Valproic Acid as an Effective Therapy for Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual.
Sponsor: CancerCare Manitoba (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Dr. David Szwajcer, Principal Investigator, CancerCare Manitoba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCM-001
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Active CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Valproic Acid; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Valproic acid & fludarabine

INTERVENTIONS:
Drug: Valproic acid & fludarabine — valproic acid (VPA) starting dose of 15 mg/day p.o. in divided doses, increased weekly by 5 mg/kg/day until >1mM Fludarabine 40 mg/m2/day orally will be added after completing 28 days of VPA if participant has been identified as having stable or progressive disease.

SUMMARY:
OBJECTIVES

To investigate:

* the mechanism of Valproic Acid (VPA)-induced apoptosis in B-CLL
* the ability of VPA in combination with standard chemotherapy or new antitumor agents to induce a synergistic antitumor effect in chronic lymphocytic leukemia (CLL) cells
* the clinical efficacy of VPA in previously treated CLL patients.

This will be an example of a translational research study where the results of our laboratory studies will be applied to a clinical trial in the CLL clinic at CancerCare Manitoba.

DETAILED DESCRIPTION:
All participants will be treated with valproic acid (VPA) at a starting dose of 15 mg/kg/day orally in divided doses. This dose produces a VPA plasma level of 346-693 μM and is the recommended starting dose for patients with seizure disorder. Each week a pre-dose serum VPA level will be determined by immunoassay and the daily dose increased by 5 mg/kg/d to ensure a predose level > 1mM. Once the target dose has been achieved serum VPA levels will be determined on a monthly basis to ensure a pre dose level >1mM.

After completing 28 days of therapy participants will be examined and have lab work drawn (CBC with differential, electrolytes, BUN, creatinine, total protein, albumin, calcium, LDH, total and direct bilirubin, ALT/AST, and β2-microglobulin. Females of child bearing age will undergo a pregnancy test prior to each 28 day cycle). For participants identified as having stable or progressive disease (National Cancer Institute Criteria), Fludarabine (Flu) therapy will be added to VPA on a 28 day cycle. Oral Flu will be administered at a dose of 40 mg/m2/day on days 1-3 of a 28 day cycle in addition to VPA as described above. Dose adjustments for Flu will be based on creatinine clearance. All participants receiving fludarabine will receive irradiated blood products and pneumocystis carnii prophylaxis.

Treatment will be continued with VPA ± Flu to a maximum of six 28 day cycles. Therapy will be discontinued prior to six 28 day cycles if: a) the participant requests discontinuation, b) if the participant is unable to comply with the protocol, c) the medical care team thinks a change of therapy would be in the best interest of the participant, d) there is evidence of progressive disease after two cycles of VPA + Flu, e) if the participant experiences unacceptable toxicity attributable to the study drugs such as ≥3 non-hematological toxicity or prolonged grade 4 hematological toxicity (NCI common toxicity criteria, Table 5 of the protocol), f) if the AST/ALT increase to > 6x the upper limit of normal or g) the participant becomes pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Active CLL (as defined by the National Cancer Institute Working Group)
* Patients must have received at least one prior therapy for CLL and have been treated with a nucleoside analogue.
* Recruitment will be limited to those with an ECOG performance status of 2 or less.

Exclusion Criteria:

* Patients who are pregnant or breastfeeding
* Patients with a history of autoimmune cytopenias
* Patients with platelets < 50 x 109/L or an absolute neutrophil count < 1.5X109/L
* Patients with hepatic disease or an AST/ALT 6x above the upper limit of normal
* Patients with a calculated creatinine clearance < 30 ml/min using the Cockroft and Gault formula
* Patients with a history of pancreatitis
* Patients who are receiving drugs that affect VPA protein binding or metabolism
* Patients with active infection, HIV or active viral hepatitis
* Patients with active secondary malignancy or who have central nervous system involvement with CLL
* Patients diagnosed with more an aggressive lymphoproliferative disorder such as Richter's transformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Best clinical response as defined by NCIWG criteria for CLL | 6 months after commencing therapy

SECONDARY OUTCOMES:
Effect of treatment on histone acetylation status; hematological toxicity (graded according to NCIWG criteria for CLL) and nonhematological toxicity (graded according to NCI common toxicity criteria) | throughout therapy

CONTACTS AND LOCATIONS:
Overall Officials: David Szwajcer, MD, Principal Investigator — CancerCare Manitoba / University of Manitoba
Locations (1):
- CancerCare Manitoba, Winnipeg, Manitoba, Canada

REFERENCES:
- See also: Official CancerCare Manitoba Website — http://cancercare.mb.ca